CLINICAL TRIAL: NCT01205620
Title: IRB-HSR# 15084 A Prospective, Unblinded, Controlled Study to Evaluate the Effect of the ITPR in Patients Undergoing OPCAB Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Responsible Party: Julie L. Huffmeyer, MD, UVA anesthehesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15084
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: CABG
Keywords: CABG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITPR (Experimental): • Upon incision of the pericardium the -9 mmHg ITPR device will be applied to the patient's endotracheal tube (in the ITPR randomized group).
  Interventions: Device: ITPR
- No intervention (No Intervention): No intervention will be performed in this control group
  Interventions: Other: No intervention

INTERVENTIONS:
Device: ITPR — • Upon incision of the pericardium the -9 mmHg ITPR device will be applied to the patient's endotracheal tube (in the ITPR randomized group).
  Arms: ITPR
Other: No intervention — No intervention will be performed in the control group
  Arms: No intervention

SUMMARY:
Participants undergoing Off-CABG will be randomized 1:1 to one of the following groups:

* treatment with CirQlator TM Intrathoracic Pressure Regulator (ITPR)
* no ITPR .Anesthesia will be standardized for both groups. The groups will be compared based on the differences in vasopressor use, the number and amount (in milliliters) of intravenous fluid boluses required and hemodynamic changes noted, including systemic blood pressure, pulmonary arterial pressure, pulse pressure, heart rate (recorded most reliably from the arterial line), cardiac output (CO), cardiac index (CI), mixed venous oxygen saturation (SVO2), SVR, pulmonary vascular resistance (PVR), and stroke volume (SV).

Specifically, we will compare the groups based on the mean number of intravenous fluid boluses, mean amount of norepinephrine and epinephrine infusion required, the number of recorded systolic blood pressures < 90 mmHg, and number of CI < 2.0 L/min/m2. We will also compare the number of times the surgeon must reposition the heart for treatment of hypotension, and ascertain whether the ITPR will help patients tolerate the cardiac displacement better, thus decreasing the time required to complete the bypass graft anastamosis. ECG will be monitored intraoperatively for signs of ischemia including ST changes, greater than 1mm depression or elevation. Postoperatively, we will record the need for and amount of diuretic required.

We hypothesize that in this pilot study, patients undergoing OPCAB who are treated with CirQlator TM Intrathoracic Pressure Regulator (ITPR) will achieve higher blood pressures and cardiac output and require less intravenous fluids and vasopressor administration than patients managed without the ITPR.

DETAILED DESCRIPTION:
A new method to improve cardiac performance during OPCAB surgery is needed in order to avoid the administration of large amounts of intravenous volume, reduce vasopressor medications, and thus improve cardiac function and reduce the need for postoperative diuresis.

The CirQlator TM Intrathoracic Pressure Regulator (ITPR) is an FDA-approved device intended to increase circulation and blood pressure in hypovolemic and cardiogenic shock. The device is inserted within a standard respiratory circuit between the patient and the ventilator. It functions by decreasing intrathoracic pressure during the expiratory phase to subatmospheric levels after each positive pressure ventilation. The decrease in intrathoracic pressure creates a vacuum within the thorax relative to the rest of the body thereby enhancing blood return to the heart and consequently increasing cardiac output and blood pressure. Activation of the device is also accompanied by a decrease in systemic vascular resistance (SVR). The end result is a device that simultaneously improves cardiac output by increasing preload and decreasing systemic vascular resistance (SVR) while increasing coronary perfusion pressure by increasing blood pressure and decreasing left ventricular end systolic pressure and volume (LVESP/LVESV).7-14

ELIGIBILITY:
Inclusion Criteria:

* patients presenting for elective off-pump CABG age 18 years of age and older informed consent has been obtained

Exclusion Criteria:

* Patients with planned on pump CABG patients requiring IABP or VAD pre-operatively emergent CABG pneumothorax hemothorax uncontrolled bleeding uncontrolled hypertension defined as SBP > 180 mmHg at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08

PRIMARY OUTCOMES:
hemodynamic changes | during surgery
  hemodynamic changes noted, including systemic blood pressure, pulmonary arterial pressure, pulse pressure, heart rate (recorded most reliably from the arterial line), cardiac output (CO), cardiac index (CI), mixed venous oxygen saturation (SVO2), SVR, pulmonary vascular resistance (PVR), and stroke volume (SV).

SECONDARY OUTCOMES:
use of vasopressors | during surgery
  the specific drug and dos will be comparedage used during surgery
IV fluids administered | during surgery
  the type & amount of fluid administered suring surgery will be compared
the number of times the surgeon must reposition the heart for treatment of hypotension | during surgery
  the number of times the surgeon must reposition the heart for treatment of hypotension will be compared, and ascertain whether the ITPR will help patients tolerate the cardiac displacement better, thus decreasing the time required to complete the bypass graft anastamosis.
cardiac ischemia | during surgery
  ECG will be monitored intraoperatively for signs of ischemia including ST changes, greater than 1mm depression or elevation.
diuretics administered | 48 hours after surgery
  Postoperatively, we will record the need for and amount of diuretic required.for the first 48 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Huffmyer, MD, Principal Investigator — UVA Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Bainbridge D, Cheng DC. Minimally invasive direct coronary artery bypass and off-pump coronary artery bypass surgery: anesthetic considerations. Anesthesiol Clin. 2008 Sep;26(3):437-52. doi: 10.1016/j.anclin.2008.03.007. PMID 18765216
- [Background] Jansen EW, Grundeman PF, Mansvelt Beck HJ, Heijmen RH, Borst C. Experimental off-pump grafting of a circumflex branch via sternotomy using a suction device. Ann Thorac Surg. 1997 Jun;63(6 Suppl):S93-6. doi: 10.1016/s0003-4975(97)00357-3. PMID 9203608
- [Background] Grundeman PF, Borst C, van Herwaarden JA, Mansvelt Beck HJ, Jansen EW. Hemodynamic changes during displacement of the beating heart by the Utrecht Octopus method. Ann Thorac Surg. 1997 Jun;63(6 Suppl):S88-92. doi: 10.1016/s0003-4975(97)00339-1. PMID 9203607
- [Background] Nierich AP, Diephuis J, Jansen EW, Borst C, Knape JT. Heart displacement during off-pump CABG: how well is it tolerated? Ann Thorac Surg. 2000 Aug;70(2):466-72. doi: 10.1016/s0003-4975(00)01561-7. PMID 10969664
- [Background] Grundeman PF. Vertical displacement of the beating heart by the Utrecht Octopus tissue stabilizer: effects on haemodynamics and coronary flow. Perfusion. 1998 Jul;13(4):229-30. doi: 10.1177/026765919801300403. No abstract available. PMID 9682254
- [Background] Grundeman PF, Borst C, Verlaan CW, Meijburg H, Moues CM, Jansen EW. Exposure of circumflex branches in the tilted, beating porcine heart: echocardiographic evidence of right ventricular deformation and the effect of right or left heart bypass. J Thorac Cardiovasc Surg. 1999 Aug;118(2):316-23. doi: 10.1016/S0022-5223(99)70222-9. PMID 10425005
- [Background] Lurie KG, Zielinski TM, McKnite SH, Idris AH, Yannopoulos D, Raedler CM, Sigurdsson G, Benditt DG, Voelckel WG. Treatment of hypotension in pigs with an inspiratory impedance threshold device: a feasibility study. Crit Care Med. 2004 Jul;32(7):1555-62. doi: 10.1097/01.ccm.0000131207.29081.a2. PMID 15241102
- [Background] Lurie KG, Zielinski T, McKnite S, Aufderheide T, Voelckel W. Use of an inspiratory impedance valve improves neurologically intact survival in a porcine model of ventricular fibrillation. Circulation. 2002 Jan 1;105(1):124-9. doi: 10.1161/hc0102.101391. PMID 11772887
- [Background] Lurie KG, Voelckel WG, Zielinski T, McKnite S, Lindstrom P, Peterson C, Wenzel V, Lindner KH, Samniah N, Benditt D. Improving standard cardiopulmonary resuscitation with an inspiratory impedance threshold valve in a porcine model of cardiac arrest. Anesth Analg. 2001 Sep;93(3):649-55. doi: 10.1097/00000539-200109000-00024. PMID 11524335
- [Background] Lurie KG, Mulligan KA, McKnite S, Detloff B, Lindstrom P, Lindner KH. Optimizing standard cardiopulmonary resuscitation with an inspiratory impedance threshold valve. Chest. 1998 Apr;113(4):1084-90. doi: 10.1378/chest.113.4.1084. PMID 9554651
- [Background] Yannopoulos D, McKnite S, Metzger A, Lurie KG. Intrathoracic pressure regulation improves 24-hour survival in a porcine model of hypovolemic shock. Anesth Analg. 2007 Jan;104(1):157-62. doi: 10.1213/01.ane.0000249047.80184.5a. PMID 17179262
- [Background] Yannopoulos D, McKnite SH, Metzger A, Lurie KG. Intrathoracic pressure regulation for intracranial pressure management in normovolemic and hypovolemic pigs. Crit Care Med. 2006 Dec;34(12 Suppl):S495-500. doi: 10.1097/01.CCM.0000246082.10422.7E. PMID 17114984
- [Background] Yannopoulos D, Metzger A, McKnite S, Nadkarni V, Aufderheide TP, Idris A, Dries D, Benditt DG, Lurie KG. Intrathoracic pressure regulation improves vital organ perfusion pressures in normovolemic and hypovolemic pigs. Resuscitation. 2006 Sep;70(3):445-53. doi: 10.1016/j.resuscitation.2006.02.005. Epub 2006 Aug 9. PMID 16901611
- [Background] Yannopoulos D, Nadkarni VM, McKnite SH, Rao A, Kruger K, Metzger A, Benditt DG, Lurie KG. Intrathoracic pressure regulator during continuous-chest-compression advanced cardiac resuscitation improves vital organ perfusion pressures in a porcine model of cardiac arrest. Circulation. 2005 Aug 9;112(6):803-11. doi: 10.1161/CIRCULATIONAHA.105.541508. Epub 2005 Aug 1. PMID 16061732